CLINICAL TRIAL: NCT02810197
Title: Etude Longitudinale En Imagerie Cérébrale, En Neuropsychologie, Et En Psychopathologie, Des Conséquences D'un Événement Traumatique
Brief Title: Resilience and Modification of Brain Control Network Following November 13
Acronym: REMEMBER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C16-13
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Neuropsychological Tests; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposed group (Experimental): Psychopathological assessment Neuropsychological assessment Functional magnetic resonance imaging (fMRI)
  Interventions: Behavioral: Psychopathological assessment; Behavioral: Neuropsychological assessment; Device: Functional magnetic resonance imaging (fMRI)
- unexposed group (Experimental): Psychopathological assessment Neuropsychological assessment Functional magnetic resonance imaging (fMRI)
  Interventions: Behavioral: Psychopathological assessment; Behavioral: Neuropsychological assessment; Device: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Behavioral: Psychopathological assessment
Behavioral: Neuropsychological assessment
Device: Functional magnetic resonance imaging (fMRI)

SUMMARY:
This is a multiwave longitudinal neuroimaging study in a cohort of direct survivors of 11/13 Paris terrorist attacks. Both structural and functional brain imaging data will be collected at 8-12 months, 3 years, and 6 years after trauma in exposed participants as well as in control non-exposed participants. This project will capitalize on recent evidence showing that healthy participants can prevent unwanted images from entering consciousness using inhibitory control and memory suppression techniques, disrupting traces of the memories in sensory areas of the brain, and weakening their vividness and later reentrance. This process is believed to be affected in Post-traumatic stress disorder (PTSD) which is characterized by anxiety and persistent intrusive memory of the traumatic event with highly distressing contents. This project will thus provide a unique opportunity to observe the online and structural dysfunctions of intrusion control network following a severe psychological trauma and how such process may contribute to recovery and psychopathological dynamics. In addition, the disruption of social cognition and emotional processing following PTSD will also be investigated in relation to disrupted inhibitory control functioning.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 and 55 years old.
* Present at the scene of the attacks the evening of 13 November 2015 or inhabitant of one of the neighbourhood affected by the attacks (exposed group), or persons were not in Paris on the evening of the attacks and not residing in Paris and its region (unexposed group).
* Affiliated to the French national health care system
* Have a good knowledge of the French language
* Right-handed
* Body mass less than or equal to 35kg/m2
* Signed written consent form

Exclusion Criteria:

* Pregnancy or intent to get pregnant
* Person deprived of their liberty
* Person admitted to a health or social institution for purposes other than research
* Minor
* Person subjected to an exclusion period related to another protocol
* History of severe psychiatric disorders before the attacks : psychotic disorders, bipolar disorder, obsessive compulsive disorder and / or substance use disorders (excluding tobacco addiction)
* Use of medication that may interfere with cognitive or cerebral functioning
* Presence of visual or hearing troubles that may compromise participant's ability to participate in the study
* MRI Contraindications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) response as measured with fMRI | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de La Sayette, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- GIP Cyceron, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coll SY, Eustache F, Doidy F, Fraisse F, Peschanski D, Dayan J, Gagnepain P, Laisney M. Avoidance behaviour generalizes to eye processing in posttraumatic stress disorder. Eur J Psychotraumatol. 2022 Apr 20;13(1):2044661. doi: 10.1080/20008198.2022.2044661. eCollection 2022. PMID 35479300